CLINICAL TRIAL: NCT00519090
Title: A Phase III Randomized, Open- Label Multi-center Study of Nilotinib Versus Imatinib in Adult Patients With Ph+ Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) Who Have a Suboptimal Cytogenetic Response (CyR) on Imatinib
Brief Title: Nilotinib vs Imatinib in Adult Patients With Philadelphia (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Acronym: ENEST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated due to limited enrollment.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2302
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Myelogenous Leukemia
Keywords: leukemia; bone marrow; leukemia symptoms; cml; complete blood count; lymphocyte; blood cancer; leukocytes; chronic leukemia; bone marrow biopsy; leukemia research; leukemia cells; bone marrow disease; chronic myeloid leukemia; blood cancer symptoms; white blood cell diseases; chronic myelogenous leukemia; leukemia treatment; leukemia facts; leucemia; facts about leukemia; myelogenous leukemia; newly diagnosed CML; suboptimal response; Philadelphia chromosome positive (Ph+); chronic myelogenous leukemia in chronic phase (CML-CP)
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hematologic Neoplasms; Bone Marrow Diseases | interventions — Imatinib Mesylate; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nilotinib (AMN107) (Experimental)
  Interventions: Drug: Nilotinib (AMN107)
- Imatinib (Active Comparator)
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Administered orally as a single agent on a continuous daily schedule given 400 mg bid (twice daily) with food. One cycle comprised of 28 days.
  Other Names: STI571; imatinib mesylate; Glivec®; Gleevec®
  Arms: Imatinib
Drug: Nilotinib (AMN107) — Administered orally as a single agent on a continuous daily schedule of 400 mg bid (2 x 200 mg twice daily) without food. Once cycle comprised of 28 days.
  Arms: Nilotinib (AMN107)

SUMMARY:
In this study, the efficacy and safety of nilotinib 400 mg twice daily, will be compared with imatinib 400 mg twice daily in patients with a suboptimal response to imatinib for their Philadelphia chromosome-positive (Ph+) Chronic Myelogenous Leukemia in the chronic phase (CML-CP).

DETAILED DESCRIPTION:
This trial was to evaluate the CCyR rate at 12 months of nilotinib therapy when compared to imatinib treatment in patients with suboptimal response to imatinib. The patients were stratified by prior duration of initial imatinib treatment, and were randomized to receive either 400 mg/twice daily of continuous nilotinib or imatinib treatment. The first stratum patients were treated with imatinib = 6 to < 12 months and having at least a minimal cytogenetic, but no partial cytogenetic response; and the second stratum patients were treated with imatinib = 12 months to < 18 months and having partial cytogenetic response (PCyR), but no CCyR.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of Philadelphia chromosome positive chronic myelogenous leukemia in the chronic phase.

Patients with suboptimal cytogenetic response to a dose of 400 mg imatinib (first line therapy) defined as:

* 6 to < 12 months of treatment and -have 36 - 95% Ph+ metaphases, or
* 12 to <18 months of treatment and have 1 - 35% Ph+ metaphases (Standard cytogenetics, no FISH [fluorescence in situ hybridization] analysis was allowed).

Exclusion criteria:

* Patient who have received more than 18 months of imatinib therapy
* Patients who have achieved partial or complete cytogenetic response and lost that response prior to entering the study.
* Prior treatment with greater than 400 mg/day imatinib.
* Uncontrolled or significant cardiovascular disease.
* Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection).
* Use of therapeutic coumarin derivatives (i.e., warfarin, acenocoumarol, phenprocoumon)
* Currently taking certain medications that could affect the rhythm of your heart.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (80):
- United States (36):
  - Arizona Cancer Center, Tucson, Arizona
  - Southern California Permanente Medical Group, Anaheim, California
  - Southern California Permanente Medical Group, Baldwin Park, California
  - Southern California Permanente Medical Group, Fontana, California
  - Kaiser Permanente Medical Group/Hayward Medical Center, Hayward, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Kaiser Permanente Medical Group/Oakland Medical Center, Oakland, California
  - Southern California Permanente Medical Group, Panorama City, California
  - Southern California Permanente Medical Group, Riverside, California
  - Kaiser Permanente Medical Group/Sacramento Medical Center, Sacramento, California
  - Southern California Permanente Medical Group, San Diego, California
  - Kaiser Permanente Medical Group, San Francisco, California
  - Kaiser Permanente Medical Group, San Jose, California
  - Kaiser Permanente Medical Group/Santa Clara Medical Office, Santa Clara, California
  - Kaiser Permanente Medical Group/South San Francisco Medical Center, South San Francisco, California
  - Kaiser Permanente Medical Group/Vallejo Medical Center, Vallejo, California
  - Kaiser Permanente Medical Group/Walnut Creek Medical Center, Walnut Creek, California
  - Southen California Permanente Medical Group, Woodland Hills, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Beech Grove, Indiana
  - Holden Cancer Center, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Methodist Cancer Center, Omaha, Nebraska
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Jones Cancer Center, Germantown, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Australia (7):
  - Novartis Investigative Site, Darlinghurst
  - Novartis Investigative Site, Herston
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Perth
  - Novartis Investigative Site, Prahran
  - Novartis Investigative Site, South Brisbane
  - Novartis Investigative Site, St Leonards
- Belgium (3):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Brazil (3):
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Porto Alegre
  - Novartis Investigative Site, São Paulo
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Germany (13):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eisensach
  - Novartis Investigative Site, Firenze
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzeg
  - Novartis Investigative Site, Postsdam
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Weiden
- Italy (6):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Reggio Calabra
  - Novartis Investigative Site, Roma
- Japan (3):
  - Novartis Investigative Site, Nagoya
  - Novartis Investigative Site, Oaska
  - Novartis Investigative Site, Tokyo
- South Korea (2):
  - Novartis Investigative Site, Hwasun-Gun
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Valencia

REFERENCES:
- [Derived] Agrawal M, Hanfstein B, Erben P, Wolf D, Ernst T, Fabarius A, Saussele S, Purkayastha D, Woodman RC, Hofmann WK, Hehlmann R, Hochhaus A, Muller MC. MDR1 expression predicts outcome of Ph+ chronic phase CML patients on second-line nilotinib therapy after imatinib failure. Leukemia. 2014 Jul;28(7):1478-85. doi: 10.1038/leu.2014.6. Epub 2014 Jan 10. PMID 24472814

RESULTS

PARTICIPANT FLOW:
Groups:
- Nilotinib (AMN107): Patients received 400 mg twice daily, 2 x 200 mg capsules twice daily.
- Imatinib: Patients received 400 mg twice daily. Capsules were available in 100 mg and 400 mg formulations.
Period: Overall Study
Arm/Group | Nilotinib (AMN107) | Imatinib
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nilotinib (AMN107) | Imatinib | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 4 | 4
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 69.5 (4.949747) | 45.5 (12.06924) | 54 (15.6812)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 0 | 1
  Germany | 0 | 1 | 1
  Japan | 1 | 0 | 1
  Korea, Republic of | 0 | 1 | 1
  Poland | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Cytogenetic Response Rate(CCyR) in Patients Who Had a Suboptimal Cytogenetic Response on Imatinib
Description: Due to early termination of the trial, the number of patients was too small and imbalanced and therefore analysis was not performed.
Time Frame: 12 months
Measure: Number; unit: percent of participants
Arm/Group | Nilotinib (AMN107) | Imatinib
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Durable Complete Cytogenetic Response Rate
Description: as for outcome 1
Time Frame: 24 months
Population: The trial was terminated early, so only 6 patients were enrolled.
Measure: Number; unit: percent of participants
Arm/Group | Nilotinib (AMN107) | Imatinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Nilotinib (AMN107) | Imatinib
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (AMN107) (N=2) | Imatinib (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Face Oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Hepatic function abnormality (Hepatobiliary disorders) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Periorbital Oedema (Eye disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Weight decrease (Metabolism and nutrition disorders) | 1 | 0
Weight increase (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data in the clinical trial.